CLINICAL TRIAL: NCT06553469
Title: Efficacy of Sacral Nerve Modulation on Urinary and Defecation Dysfunction After Spinal Cord Injury
Brief Title: Efficacy of Sacral Nerve Modulation on Urinary and Defecation Dysfunction After Spinal Cord Injury：A Prospective, Single-arm Study
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: YL01
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Cystometry; Sacral Neuromodulation; Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SNM group: After screening according to the inclusion and exclusion criteria, the subjects were enrolled in the study. The sacral nerve regulation treatment was divided into two phases. Phase I was the testing phase, during which sacral nerve stimulation electrode component implantation was performed. After electrode implantation, testing was conducted for 2-4 weeks. According to the urine diary and scale scores, if the symptoms improved by ≥ 50%, or if the patient requested to continue with phase II and was evaluated by the researcher as suitable for implantation, phase II (permanent implantation phase) treatment was performed, and sacral nerve stimulation pulse generator component implantation was performed.During the trial period, all patients in the intervention group received routine care for neurogenic lower urinary tract dysfunction, including regular clean interval catheterization (CIC), in addition to sacral nerve regulation therapy
  Interventions: Device: sacral neuromodulation

INTERVENTIONS:
Device: sacral neuromodulation — After screening according to the inclusion and exclusion criteria, the subjects were enrolled in the study. The sacral nerve regulation treatment was divided into two phases. Phase I was the testing phase, during which the sacral nerve stimulation electrode component was implanted. After the electrode was implanted, it was tested for 2-4 weeks. According to the urine diary and scale scores, if the symptoms improved by ≥ 50%, or if the patient requested to continue with Phase II and was evaluated by the researcher as suitable for implantation, Phase II (permanent implantation phase) treatment was performed, during which the sacral nerve stimulation pulse generator component was implanted

SUMMARY:
The aim of this study is to investigate the long-term efficacy of sacral nerve modulation surgery in the treatment of neurogenic lower urinary tract dysfunction caused by incomplete spinal cord injury, as well as its preventive effect on complications of neurogenic lower urinary tract dysfunction. We will use urodynamic examination results such as maximum bladder capacity and detrusor leak point pressure, combined with renal function and urinary ultrasound results, as our evaluation indicators. Follow up evaluations will be conducted at 6 and 12 months after permanent implantation, and periodic comparisons will be made with baseline data to gain a more comprehensive understanding of the effectiveness and safety of sacral nerve regulation surgery.

DETAILED DESCRIPTION:
Spinal cord injury is a serious type of central nervous system injury that not only causes movement disorders, but also damages the bladder, intestines, and autonomic nervous circuits related to sexual function, leading to urinary and defecation disorders. Sacral nerve modulation is a technology that applies low-frequency electric pulse to specific sacral nerve continuously to affect and regulate the function of target organs, so as to treat urgent urinary incontinence, overactivity of bladder, urinary retention, fecal incontinence and other diseases. However, there is currently no consensus on whether this technology can treat urinary and defecation dysfunction caused by spinal cord injury, and its specific mechanism still needs to be studied. Existing research shows that this technique can reduce the excitability of sphincter by inhibiting the protective reflex to treat urinary retention; Treating detrusor overactivity by inhibiting detrusor muscle activity without affecting urethral resistance and detrusor muscle contraction during urination. This study hypothesizes that sacral nerve modulation intervention after spinal cord injury can reduce bladder spasms, maintain bladder compliance, bladder capacity, and low bladder filling pressure, delay the progression of bladder fibrosis and hydronephrosis after spinal cord injury, and improve symptoms such as constipation. Based on the above evidence and hypotheses, we designed a single arm clinical trial to evaluate the effectiveness and safety of sacral nerve modulation surgery in treating urinary and defecation dysfunction after incomplete spinal cord injury, especially in preventing complications such as bladder fibrosis and hydronephrosis. We also evaluated the impact of sacral nerve modulation surgery on the quality of life of patients after spinal cord injury, as well as the improvement effect of sacral nerve modulation surgery on urinary and reproductive system related symptoms and intestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old, gender not limited
* Diagnosed with urinary and defecation dysfunction caused by spinal cord injury
* Urodynamic examination suggests bladder dysfunction
* ASIA spinal cord injury classification: B, C, or D
* Safe bladder capacity>100ml
* Patients who can undergo sacral nerve regulation surgery after evaluation
* If you plan not to combine medication during the study period, you need to stop taking the medication for at least 7 days before the screening period. If you plan to continue drug treatment during the study period, you need to maintain the same dosage or stop taking the medication after evaluation by a doctor.
* Voluntarily participate in this clinical study, and the subjects sign a written informed consent form before the start of the study.
* After testing treatment, if any of the following conditions are met, permanent implantation of a sacral nerve stimulator is feasible① The average daily frequency of urination during the last 3 days of experiential therapy decreased by ≥ 50% compared to baseline;② The average urinary urgency score for the last 3 days of experiential therapy decreased by ≥ 50% compared to baseline; ③ The number of urinary incontinence episodes in the last 3 days of experiential therapy decreased by ≥ 50% compared to baseline;④ The average urine output per session during the last 3 days of experiential therapy increased by ≥ 50% compared to baseline;⑤ The patient requires permanent implantation due to improvement in intestinal and sexual function, and after evaluation by the researcher, can undergo phase II treatment

Exclusion Criteria:

* Other causes of lower urinary tract dysfunction cannot be ruled out, or other diseases that may lead to lower urinary tract dysfunction cannot be ruled out
* Pregnant women, lactating women, women of childbearing age who plan to conceive or have no safe contraceptive measures during the study period
* Patients with mental and cognitive impairments, as well as those who are unable to cooperate with the experimental process
* Patients with untreated infections, coagulation disorders, malignant tumors, and other serious illnesses
* Individuals who have undergone other relevant surgical treatments within 3 months prior to enrollment (including but not limited to bladder wall injection of botulinum toxin type A), or have participated in other clinical trials
* Other situations that researchers consider inappropriate to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects were patients from Qilu Hospital, Shandong University.Recruitment process for research subjects:(1) Preliminary screening of patients based on admission and exclusion criteria;(2) Promote clinical trials to potential participants;(3) The assistant shall compile and organize the basic information and intention to participate in the trial of personnel who meet the recruitment requirements, inform them of the procedures for participating in the trial, and arrange for the recruitment of candidates to participate in the trial screening;(4) Researchers will further screen the recruited subjects according to the requirements of the experimental plan, and those who meet the requirements will be assigned to the group and included in the normal experimental procedure; For those that do not meet the requirements, notify the assistant to handle subsequent matters, such as explaining the work, distributing transportation subsidies, etc
Sampling Method: Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
urodynamics | 3,6,12 month
  To examine function of bladder
renal function | 3,6,12 month
  To examine function of kidney
Urinary ultrasound | 3,6,12 month
  morphological change of urinary system

CONTACTS AND LOCATIONS:
Overall Officials: Lipeng Chen, Dortor, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jazayeri SB, Maroufi SF, Mohammadi E, Dabbagh Ohadi MA, Hagen EM, Chalangari M, Jazayeri SB, Safdarian M, Zadegan SA, Ghodsi Z, Rahimi-Movaghar V. Incidence of traumatic spinal cord injury worldwide: A systematic review, data integration, and update. World Neurosurg X. 2023 Feb 1;18:100171. doi: 10.1016/j.wnsx.2023.100171. eCollection 2023 Apr. PMID 36910686
- [Background] Quadri SA, Farooqui M, Ikram A, Zafar A, Khan MA, Suriya SS, Claus CF, Fiani B, Rahman M, Ramachandran A, Armstrong IIT, Taqi MA, Mortazavi MM. Recent update on basic mechanisms of spinal cord injury. Neurosurg Rev. 2020 Apr;43(2):425-441. doi: 10.1007/s10143-018-1008-3. Epub 2018 Jul 11. PMID 29998371
- [Background] Redshaw JD, Lenherr SM, Elliott SP, Stoffel JT, Rosenbluth JP, Presson AP, Myers JB; Neurogenic Bladder Research Group (NBRG.org). Protocol for a randomized clinical trial investigating early sacral nerve stimulation as an adjunct to standard neurogenic bladder management following acute spinal cord injury. BMC Urol. 2018 Aug 29;18(1):72. doi: 10.1186/s12894-018-0383-y. PMID 30157824